CLINICAL TRIAL: NCT02893371
Title: Longitudinal Comparative Effectiveness of Bipolar Disorder Therapies
Status: Terminated | Type: Observational
Why Stopped: Per PI, this study is not a clinical trial and was inadvertently entered in the system
Sponsor: University of New Mexico (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Montana State University (Other); National Alliance on Mental Illness Montana (Unknown); CGStat LLC (Other); Risk Benefit Statistics LLC (Industry); National Alliance on Mental Illness New Mexico (Unknown); National Alliance on Mental Illness Westside Los Angeles (Unknown)
Responsible Party: Principal Investigator, Christophe Gerard Lambert, Associate Professor, University of New Mexico
Other Study IDs: 16-243; CER-1507-31607 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium Carbonate; Lamotrigine; Valproic Acid; Oxcarbazepine; Carbamazepine; ziprasidone; Risperidone; Quetiapine Fumarate; Olanzapine; Aripiprazole; olanzapine-fluoxetine combination; Haloperidol; Perphenazine; Clozapine; asenapine; Lurasidone Hydrochloride; Paliperidone Palmitate; Mirtazapine; Bupropion; Desvenlafaxine Succinate; Duloxetine Hydrochloride; Venlafaxine Hydrochloride; Citalopram; Escitalopram; Fluoxetine; Fluvoxamine; Paroxetine; Sertraline; Vilazodone Hydrochloride; Doxepin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lithium Carbonate — Exposure to all dosages and delivery forms.
  Other Names: Lithobid
Drug: Lamotrigine — Exposure to all dosages and delivery forms.
  Other Names: Lamictal
Drug: Valproic Acid — Exposure to all dosages and delivery forms.
  Other Names: Depakote; Valproate
Drug: Oxcarbazepine — Exposure to all dosages and delivery forms.
  Other Names: Trileptal
Drug: Carbamazepine — Exposure to all dosages and delivery forms.
  Other Names: Equetro
Drug: Ziprasidone — Exposure to all dosages and delivery forms.
  Other Names: Geodon
Drug: Risperidone — Exposure to all dosages and delivery forms.
  Other Names: Risperdal
Drug: Quetiapine — Exposure to all dosages and delivery forms.
  Other Names: Seroquel
Drug: Olanzapine — Exposure to all dosages and delivery forms.
  Other Names: Zyprexa
Drug: Aripiprazole — Exposure to all dosages and delivery forms.
  Other Names: Abilify
Drug: Fluoxetine / Olanzapine — Exposure to all dosages and delivery forms.
  Other Names: Symbyax
Drug: Haloperidol — Exposure to all dosages and delivery forms.
  Other Names: Haldol Decanoate
Drug: Perphenazine — Exposure to all dosages and delivery forms.
  Other Names: Trilafon
Drug: Clozapine — Exposure to all dosages and delivery forms.
  Other Names: Clozaril
Drug: Asenapine — Exposure to all dosages and delivery forms.
  Other Names: Saphris
Drug: Lurasidone — Exposure to all dosages and delivery forms.
  Other Names: Latuda
Drug: Paliperidone — Exposure to all dosages and delivery forms.
  Other Names: Invega
Drug: Mirtazapine — Exposure to all dosages and delivery forms.
  Other Names: Remeron; Remeronsoltab
Drug: Bupropion — Exposure to all dosages and delivery forms.
  Other Names: Zyban; Aplenzin; Wellbutrin
Drug: Desvenlafaxine — Exposure to all dosages and delivery forms.
  Other Names: Pristiq; Desfax
Drug: Duloxetine — Exposure to all dosages and delivery forms.
  Other Names: Cymbalta; Irenka
Drug: Venlafaxine — Exposure to all dosages and delivery forms.
  Other Names: Effexor XR
Drug: Citalopram — Exposure to all dosages and delivery forms.
  Other Names: Celexa
Drug: Escitalopram — Exposure to all dosages and delivery forms.
  Other Names: Lexapro
Drug: Fluoxetine — Exposure to all dosages and delivery forms.
  Other Names: Prozac; Sarafem
Drug: Fluvoxamine — Exposure to all dosages and delivery forms.
  Other Names: Faverin; Fevarin; Floxyfral; Dumyrox; Luvox
Drug: Paroxetine — Exposure to all dosages and delivery forms.
  Other Names: Paxil; Seroxat
Drug: Sertraline — Exposure to all dosages and delivery forms.
  Other Names: Zoloft
Drug: Vilazodone — Exposure to all dosages and delivery forms.
  Other Names: Viibryd
Drug: Doxepin — Exposure to all dosages and delivery forms.
  Other Names: Sinequan; Silenor

SUMMARY:
The objective of this retrospective observational study is to compare commonly prescribed bipolar disorder medications for their impact on: (1) hospitalization; (2) suicide attempts and self-harm; and (3) risk of drug-induced adverse effects such as kidney disease and diabetes mellitus. In addition, the investigators will examine heterogeneity of treatment effect by co-morbidity within pediatric, adult, and elderly sub-populations. Patient focus groups are convened to elicit additional questions and provide feedback on results.

DETAILED DESCRIPTION:
Funded by PCORI, the objective of this retrospective observational study is to perform several safety and effectiveness comparisons on commonly prescribed bipolar disorder medications, engaging patient focus groups in generating additional questions and interpreting results.

The study will be a retrospective cohort study conducted with administrative claims data from the Truven MarketScan Commerical Claims and Encounters and Medicare database from 2010-2016.

The database contains approximately 140 million patients within the US population in every state and nearly every county in the nation, across all ages, ethnicities and socioeconomic categories, including privately insured, and Medicare patients. The study will focus on approximately one million patients with two or more diagnoses of bipolar disorder in the claims records according to ICD-9 and/or ICD-10 coding.

The treatments that will be compared are lithium carbonate; first generation antipsychotics: haloperidol and perphenazine; second generation antipsychotics: clozapine, risperidone, olanzapine, aripiprazole, quetiapine, ziprasidone, asenapine, lurasidone, and paliperidone; mood stabilizing anticonvulsants: valproate, lamotrigine, carbamazepine, and oxcarbazepine; antidepressants: mirtazapine, bupropion, desvenlafaxine, duloxetine, venlafaxine, citalopram, escitalopram, fluoxetine, fluvoxamine, paroxetine, sertraline, vilazodone, and doxepin.

The investigators will perform cross-sectional and survival based analysis using regression, propensity scoring, and local control to perform bias-corrected comparisons of the above treatments for for their impact on: (1) hospitalization; (2) suicide attempts and self-harm; and (3) risk of drug-induced adverse effects such as kidney disease and diabetes mellitus. In addition, the investigators will examine heterogeneity of treatment effect by co-morbidity within pediatric, adult, and elderly sub-populations.

ELIGIBILITY:
Inclusion Criteria:

* Two or more instances of bipolar disorder diagnoses within administrative claims records

Exclusion Criteria:

* Patients with less than 1 year of history in the database

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of individuals with bipolar disorder enrolled with private insurers or with Medicare across the United States, as captured in the Truven Health Analytics MarketScan databases. The time period of data coverage is 2003-2016.
Sampling Method: Non-Probability Sample
Enrollment: 1037352 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Risk of hospitalization | 0-7 years
  For each treatment, assess the risk of rehospitalization within 30-days after hospitalization for a mood episode. For each treatment, assess the cumulative incidence of hospitalization for a mood episode any time after commencing treatment, accounting for the competing risk of ending treatment.
Risk of suicide and self-harm | 0-7 years
  For each treatment, assess the cumulative risk of a second suicide or self-harm event after diagnosis of a first event, accounting for the competing risk of ending treatment. Self-harm includes injuries of unknown intent.

SECONDARY OUTCOMES:
Kidney disease | 0-7 years
  For each treatment, assess time to first instance of renal condition.
Diabetes mellitus | 0-7 years
  For each treatment, assess time to diagnosis of diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Christophe G Lambert, PhD, Principal Investigator — University of New Mexico Health Sciences Center
Locations (1):
- Christophe G Lambert, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
This retrospective observational study makes use of MarketScan individual level patient data from Truven Health Analytics. The license terms for data access prohibit public dissemination of individual level patient data. The investigators will, however, make openly available the queries and analytic procedures required to reproduce the study.

REFERENCES:
- [Result] Nestsiarovich A, Hurwitz NG, Nelson SJ, Crisanti AS, Kerner B, Kuntz MJ, Smith AN, Volesky E, Schroeter QL, DeShaw JL, Young SS, Obenchain RL, Krall RL, Jordan K, Fawcett J, Tohen M, Perkins DJ, Lambert CG. Systemic challenges in bipolar disorder management: A patient-centered approach. Bipolar Disord. 2017 Dec;19(8):676-688. doi: 10.1111/bdi.12547. Epub 2017 Sep 13. PMID 28901625
- [Result] Nestsiarovich A, Mazurie AJ, Hurwitz NG, Kerner B, Nelson SJ, Crisanti AS, Tohen M, Krall RL, Perkins DJ, Lambert CG. Comprehensive comparison of monotherapies for psychiatric hospitalization risk in bipolar disorders. Bipolar Disord. 2018 Dec;20(8):761-771. doi: 10.1111/bdi.12665. Epub 2018 Jun 19. PMID 29920885
- [Result] Nestsiarovich A, Kerner B, Mazurie AJ, Cannon DC, Hurwitz NG, Zhu Y, Nelson SJ, Oprea TI, Unruh ML, Crisanti AS, Tohen M, Perkins DJ, Lambert CG. Comparison of 71 bipolar disorder pharmacotherapies for kidney disorder risk: The potential hazards of polypharmacy. J Affect Disord. 2019 Jun 1;252:201-211. doi: 10.1016/j.jad.2019.04.009. Epub 2019 Apr 8. PMID 30986735
- [Result] Kerner B, Crisanti AS, DeShaw JL, Ho JG, Jordan K, Krall RL, Kuntz MJ, Mazurie AJ, Nestsiarovich A, Perkins DJ, Schroeter QL, Smith AN, Tohen M, Volesky E, Zhu Y, Lambert CG. Preferences of Information Dissemination on Treatment for Bipolar Disorder: Patient-Centered Focus Group Study. JMIR Ment Health. 2019 Jun 25;6(6):e12848. doi: 10.2196/12848. PMID 31237566
- [Result] Kumar P, Nestsiarovich A, Nelson SJ, Kerner B, Perkins DJ, Lambert CG. Imputation and characterization of uncoded self-harm in major mental illness using machine learning. J Am Med Inform Assoc. 2020 Jan 1;27(1):136-146. doi: 10.1093/jamia/ocz173. PMID 31651956
- [Result] Nestsiarovich A, Kerner B, Mazurie AJ, Cannon DC, Hurwitz NG, Zhu Y, Nelson SJ, Oprea TI, Crisanti AS, Tohen M, Perkins DJ, Lambert CG. Diabetes mellitus risk for 102 drugs and drug combinations used in patients with bipolar disorder. Psychoneuroendocrinology. 2020 Feb;112:104511. doi: 10.1016/j.psyneuen.2019.104511. Epub 2019 Nov 9. PMID 31744781
- [Result] Nestsiarovich A, Kumar P, Lauve NR, Hurwitz NG, Mazurie AJ, Cannon DC, Zhu Y, Nelson SJ, Crisanti AS, Kerner B, Tohen M, Perkins DJ, Lambert CG. Using Machine Learning Imputed Outcomes to Assess Drug-Dependent Risk of Self-Harm in Patients with Bipolar Disorder: A Comparative Effectiveness Study. JMIR Ment Health. 2021 Apr 21;8(4):e24522. doi: 10.2196/24522. PMID 33688834